CLINICAL TRIAL: NCT04581655
Title: Retrospective and Prospective Analysis of Risk and Outcome Factors in Oncohematological Patients Admitted to Italian Pediatric Intensive Care Units: a Multicenter Study
Brief Title: ONCOTIPNET: Multicenter Study on Risk Factors and Outcome in Cancer Pediatric Patients Admitted in Italian PICUs
Acronym: ONCOTIPNET
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: ONCOTIPNET
Record Dates: First submitted 2020-09-21; First posted 2020-10-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Cancer; Critically Ill
Keywords: pediatric intensive care unit; oncology
MeSH Terms: conditions — Neoplasms; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will describe characteristics of pediatric cancer patients admitted to Italian PICUs and will analyze risk factors of PICU admission, neurological outcome, and mortality. After a retrospective analysis (2019-2020), investigators will perform a prospective study over 12 months gathering data from 15-20 Italian PICUs.

DETAILED DESCRIPTION:
The study aim to evaluate:

1. characteristics of pediatric cancer patients admitted to Italian PICUs
2. risk factors of PICU admission, neurological outcome and mortality.

Inclusion criteria: age <= 18 years, informed consent. Exclusion criteria: informed consent not obtained. After a retrospective analysis (2019-2020), investigators will perform a prospective study over 12 months (March 2021 - February 2021) gathering data from 15-20 Italian PICUs. Each Center can decide whether to participate only in the prospective phase. Data will be recorded in an electronic data collection form in Red Cap.

The following variables will be collected:

* Demographic variables: age, sex, ethnicity;
* TIP pre-admission clinical variables and at the time of admission: basic diagnosis, comorbidity, Hemopoietic Stem Cell Transplantation (TCSE) number and type, treatment phase, HLA matching, Graft Versus Host (GVH) and grade, veno-occlusive disease, Venous Occlusive Disease
* Variables upon entering TIP: PIM3, POPC score, organ failure cause and staging, high intensity treatments, high flow oxygen therapy, dialysis, inotropes or other, fluid overload, immunodeficiency
* Clinical variables during hospitalization: organ failure cause and staging, ventilation, modality, presence of pARDS and severity, need for inotropic support, sepsis and severity score (SOFA), inotropes (VIS score), arrest event cardiac, need for HFOV, Extra-Corporeal Membrane Oxygenator, Nitric Oxide, dialysis, Intracranial Pressure monitoring, drugs used for sedation, development of withdrawal syndrome, development of delirium.

Considering the participation of 15-20 centers involving 20 patients in a year, the expected number is 600 patients considering the retrospective phase (optional, therefore some Centers may not contribute) and the prospective phase.

Study sites will also take part to a survey designed to collect data in order to describe Italian PICUs involved in providing care to cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age <= 18 yeras
* informed consent*

Exclusion Criteria:

* informed consent not obtained*

  * only for next prospective part of the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with cancer disease admitted in PICU
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
mortality | from date of patient's admission in PICU to date of PICU discharge assessed up to 7 days
  rate of dead patients
mortality | from discharge to 30th day after PICU discharge
  30-days mortality
mortality | from 31st to 90th day after PICU discharge
  90-days mortality
neurological outcome | on date of PICU discharge assessed up to 10 days
  patients's Pediatric Overall Performance Category (POPC) score (a 6 level score: 4 to 6 is considered bad outcome)

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, Dr, Principal Investigator — University Hospital Padova
Locations (17):
- Italy (17):
  - Salesi Hospital, Ancona
  - Giovanni XIII Hospital, Bergamo
  - University Hospital Policlinico S.Orsola-IRCCS, Bologna
  - Spedali Civili Hospital, University of Brescia, Brescia
  - I Policlinico, Catania
  - Meyer Hospital, Florence
  - Gaslini Hospital, Genova
  - University of Messina, Messina
  - Children's Hospital V. Buzzi-Sacco, Milan
  - Santobono Hospital, Napoli
  - Azienda Ospedale Università Padova, Padua
  - Di Cristina Hospital, Palermo
  - "Bambino Gesù" Children's Hospital, Roma
  - Regina Margherita Hospital, Torino
  - Burlo Garofalo Hospital, Trieste
  - University Hospital, Verona, Verona
  - S.Bortolo Hospital, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided
We will share individual participant data set with participating centers. Moreover we will share: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR)

REFERENCES:
- [Result] Pillon M, Amigoni A, Contin A, Cattelan M, Carraro E, Campagnano E, Tumino M, Calore E, Marzollo A, Mainardi C, Boaro MP, Nizzero M, Pettenazzo A, Basso G, Messina C. Risk Factors and Outcomes Related to Pediatric Intensive Care Unit Admission after Hematopoietic Stem Cell Transplantation: A Single-Center Experience. Biol Blood Marrow Transplant. 2017 Aug;23(8):1335-1341. doi: 10.1016/j.bbmt.2017.04.016. Epub 2017 Apr 28. PMID 28461212
- [Result] Pillon M, Sperotto F, Zattarin E, Cattelan M, Carraro E, Contin AE, Massano D, Pece F, Putti MC, Messina C, Pettenazzo A, Amigoni A. Predictors of mortality after admission to pediatric intensive care unit in oncohematologic patients without history of hematopoietic stem cell transplantation: A single-center experience. Pediatr Blood Cancer. 2019 Oct;66(10):e27892. doi: 10.1002/pbc.27892. Epub 2019 Jun 28. PMID 31250548
- [Result] Wosten-van Asperen RM, van Gestel JPJ, van Grotel M, Tschiedel E, Dohna-Schwake C, Valla FV, Willems J, Angaard Nielsen JS, Krause MF, Potratz J, van den Heuvel-Eibrink MM, Brierley J; POKER (PICU Oncology Kids in Europe Research group) research consortium. PICU mortality of children with cancer admitted to pediatric intensive care unit a systematic review and meta-analysis. Crit Rev Oncol Hematol. 2019 Oct;142:153-163. doi: 10.1016/j.critrevonc.2019.07.014. Epub 2019 Aug 3. PMID 31404827
- [Result] Faraci M, Bagnasco F, Giardino S, Conte M, Micalizzi C, Castagnola E, Lampugnani E, Moscatelli A, Franceschi A, Carcillo JA, Haupt R. Intensive care unit admission in children with malignant or nonmalignant disease: incidence, outcome, and prognostic factors: a single-center experience. J Pediatr Hematol Oncol. 2014 Oct;36(7):e403-9. doi: 10.1097/MPH.0000000000000048. PMID 24276033
- [Derived] Amigoni A, Boscato S, Mondardini MC, Cavagnero F, Marchetto L, Biassoni V, Birolo C, Bottari G, Corno M, Ferrario S, Maiolo G, Montaguti A, Rossetti E, Rulli I, Sagredini R, Spaggiari S, Vatiero L, Vigna G, Martinato M, Gregori D, Pillon M, Comoretto RI; OncoTIPNet Study Group. Exploring risk factors for pediatric cancer patients admitted to the Pediatric Intensive Care Unit: insight from a multicenter observational study revealing no association with mechanical ventilation. J Anesth Analg Crit Care. 2025 Oct 14;5(1):63. doi: 10.1186/s44158-025-00275-6. PMID 41088488